CLINICAL TRIAL: NCT01610765
Title: A Safety and Dose-Determining Study of CMX001 In Infants With Neonatal Herpes Simplex Virus (HSV) Infection Involving the Central Nervous System (CNS Disease)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated because unable to obtain access to study drug for study population.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Kimberlin, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMID 11-0068
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Herpes Simplex Virus
Keywords: HSV; pharmacokinetics; herpes; neonates
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Novel Antiviral Drug (Active Comparator): Subjects will be randomized to receive one of 3 oral doses of a Novel Antiviral Drug: 0.50 mg/kg/dose, 1.0 mg/kg/dose or 2.0 mg/kg/dose twice a week for up to 3 weeks during the time in which the 21 day administration of parenteral acyclovir is being administered
  Interventions: Drug: Novel Antiviral Drug
- Placebo (Placebo Comparator): Subjects will be randomized to receive one of 3 oral doses of placebo matched in volume to active drug: 0.50 mg/kg/dose, 1.0 mg/kg/dose or 2.0 mg/kg/dose twice a week for up to 3 weeks during the time in which the 21 day administration of parenteral acyclovir is being administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Novel Antiviral Drug — 4 oral doses of a Novel Antiviral Drug: 0.25 mg/kg/dose, 0.50 mg/kg/dose, 1.0 mg/kg/dose or 2.0 mg/kg/dose twice a week for 3 weeks during the time in which the 21 day administration of parenteral acyclovir is being administered. Subjects will be assigned a the higher dose of study drug after the DSMB and sponsor determine that reported adverse events and the PK data show that it is safe to increase dosing to the next higher level.
  Arms: Novel Antiviral Drug
Drug: Placebo — 4 oral doses of placebo matching the a Novel Antiviral Drug assigned dose: 0.25 mg/kg/dose, 0.50 mg/kg/dose, 1.0 mg/kg/dose or 2.0 mg/kg/dose twice a week for 3 weeks during the time in which the 21 day administration of parenteral acyclovir is being administered. Subjects will be assigned a the higher dose of study drug after the DSMB and sponsor determine that reported adverse events and the PK data show that it is safe to increase dosing to the next higher level.
  Arms: Placebo

SUMMARY:
This study is to identify if a Novel Antiviral Drug could be used to treat babies with Herpes Simplex Virus (HSV) with central nervous system (CNS) disease. In this study the investigators will identify the best dose for young children as well as identify additional safety information about the Novel Antiviral Drug.

DETAILED DESCRIPTION:
In this study, the pharmacokinetics and safety of a Novel Antiviral Drug will be determined in babies with neonatal HSV CNS disease. The study will be conducted at 18 academic medical centers throughout the United States. Young infants presenting with virologic confirmation of neonatal HSV infection and evidence of CNS involvement will be eligible for study enrollment. Study Day 1 is defined as the day when dose 1 of the Novel Antiviral Drug study medication is administered.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent by parent or legal guardian of study subject
* Virologically confirmed HSV infection [e.g., positive culture, DNA detection by polymerase chain reaction (PCR), or direct fluorescent antibody stain from any body site or compartment]
* Evidence of CNS involvement of HSV disease [e.g., CSF pleocytosis, positive CSF PCR testing, clinical or electroencephalogram (EEG) seizure activity, neuroimaging abnormality)
* Starting parenteral acyclovir therapy at time of initiation of CMX001 study drug or receiving parenteral acyclovir therapy for ≤ 72 hours before start CMX001 study drug
* ≤ 6 weeks (42 days) of age at time of initial onset of disease symptoms or signs
* Weight at study enrollment ≥ 2,630 grams
* Gestational age ≥ 36 weeks at delivery
* Mother tested negative for HIV during or following pregnancy

Exclusion Criteria:

* Imminent demise
* Disseminated or skin/eye/mouth (SEM) neonatal HSV disease classifications
* Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., history of necrotizing enterocolitis, gastroschisis, malrotation, etc.)
* Birth weight < 2,500 grams
* Birth weight > 4,500 grams
* Grade 3 or 4 vomiting, utilizing the DAIDS Toxicity Tables (Appendix B)
* Grade 3 or 4 diarrhea, utilizing the DAIDS Toxicity Tables (Appendix B)
* Creatinine clearance < 15 mL/min/1.73m2
* Serum albumin < 2.0 g/dL
* Alanine aminotransferase (ALT) ≥ 2.6-times upper limit normal (ULN)
* Aspartate aminotransferase (AST) ≥ 2.6-times upper limit normal (ULN)
* Direct bilirubin > 2 mg/dL
* Known immunodeficiency
* Known congenital infection (e.g., symptomatic congenital cytomegalovirus infection; syphilis; congenital toxoplasmosis)
* Congenital heart disease (e.g., patent ductus arteriosus, Tetralogy of Fallot, hypoplastic left heart syndrome, AV canal, VSD, ASD, transposition of the great arteries, hypoplastic right ventricle, truncus arteriosus, pulmonic stenosis, Ebstein anomaly, coarctation of the aorta, interrupted aortic arch, double outlet right ventricle, dilated cardiomyopathy)
* Infants currently receiving or anticipated to need treatment with digoxin that cannot be withheld for the duration of CMX001 therapy
* Infants currently receiving or anticipated to need treatment with ketaconazole that cannot be withheld for the duration of CMX001 therapy
* Receipt of investigation drugs within 30 days prior to enrollment
* Concurrent enrollment or participation in any other interventional research study

Ages: 1 Day to 98 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of CMX001 oral suspension in infants being treated for neonatal HSV CNS disease. | Baseline through day 21
Determine the plasma pharmacokinetics of the CMX001 and cidofovir following administration of CMX001 oral suspension in infants being treated for neonatal HSV CNS disease. | Baseline through day 21

SECONDARY OUTCOMES:
Explore a plasma drug concentration-response relationship between CMX001 exposure and quantity of HSV DNA in cerebrospinal fluid (CSF) at Day 4 of antiviral therapy | Baseline through day 21
Explore a plasma drug concentration-response relationship between cidofovir exposure and quantity of HSV DNA in cerebrospinal fluid (CSF) at Day 4 of antiviral therapy | Baseline through day 56 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: David W Kimberlin, MD, Principal Investigator — University of Alabama at Birmingham; Richard Whitley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Colorado at Denver Health Sciences Center, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of South Florida School of Medicine, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Louisiana State University Health Science Center -Shreveport, Shreveport, Louisiana
  - Washington University in St Louis School of Medicine, St Louis, Missouri
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Steven & Alexandra Cohen Children's Medical Center Of New York (CCMC), Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Medical Center - Charlotte, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas-Southwestern, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah